CLINICAL TRIAL: NCT03430115
Title: Long-term Function and Health Effects of Intentional Weight Loss in Obese Elders
Brief Title: Health Outcomes After Participating in Exercise (HOPE)
Acronym: HOPE
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00043576; 1R01AG056418-01 (NIH)
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Weight Loss; Obesity; Aging
Keywords: Obese; Exercise
MeSH Terms: conditions — Weight Loss; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum, plasma, PBMCs
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Weight loss plus exercise (WL+EX): This group was randomized and previously assigned to weight loss plus exercise.
- Exercise alone (EX): This group was randomized and previously assigned to exercise alone.
- Weight loss alone (WL): This group was randomized and previously assigned to weight loss alone.
- Control: This group was randomized and previously assigned to control.

SUMMARY:
Aging is associated with significant declines in muscle mass, strength, and physical performance, all of which lead to disability, loss of independence, and adverse clinical outcomes. Obesity exacerbates these age-related declines in function and is associated with poorer clinical outcomes and quality of life. Weight loss can also worsen age-related loss of muscle mass and decrease bone mineral density. The overall goals of this study are to determine if the short-term functional benefits of intentional weight loss are sustained long-term, and to examine the long-term benefits and risks of weight loss.

DETAILED DESCRIPTION:
Obesity exacerbates age-related declines in function and is associated with poorer clinical outcomes and quality of life. Although clinical trials conducted study teams show that diet-induced weight loss interventions in obese older adults, when combined with exercise, improve body composition and physical and metabolic function in the short-term, the overall safety and long-term benefits of intentional weight loss in older adults remain controversial. Weight loss can also worsen age-related loss of muscle mass and decrease bone mineral density. Because of these concerns, health care providers are reluctant to recommend weight loss in obese older adults. The goal is to determine whether weight loss-induced improvements in body composition and physical and metabolic function observed in short-term clinical trials persist over time is critical to inform geriatric obesity treatment.

ELIGIBILITY:
Inclusion Criteria:

* All former participants from the five intervention trials who respond to our recruitment strategies will be scheduled for clinic/home visits or a phone interview.

Exclusion Criteria:

* None - all former participants from the five intervention trials are eligible

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants aged 60 and older at randomization who were randomized to a weight loss intervention that was combined with an exercise intervention (WL+EX, n=392), to an exercise intervention alone (EX alone, n=340), to a weight loss intervention alone (n=128), or to a control group (n=106) from five weight loss and exercise randomized controlled trials.
Sampling Method: Non-Probability Sample
Enrollment: 588 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2021-07-27 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
400 meter walk time | Baseline
  Participants are instructed to complete the 400 m distance (on a flat indoor surface) as quickly as possible at a maintainable pace and the time to complete the walk is recorded in seconds.

SECONDARY OUTCOMES:
Short Physical Performance Battery score | Baseline
  The Short Physical Performance Battery (SPPB) is a widely used assessment of lower extremity physical function that consists of 3 standing balance tasks held for 10 seconds each (side-by-side, tandem and semi-tandem), two 4-m walk tests to assess usual gait speed, and 5 repeated chair stands. Each of the three performance measures is assigned a score ranging from 0 (inability to do the test) to 4 (the highest level of performance) and summed to create an SPPB summary score ranging from 0 (worst) to 12 (best).
Knee extension strength | Baseline
  Maximal isokinetic knee extension strength. Maximal isokinetic knee extension strength will be measured using an isokinetic dynamometer (Biodex) at 60°/sec with the participant sitting and the hips and knee flexed at 90°. The maximum knee extensor strength of the 4 repetitions from trial 2 for the dominant leg will be will be used in analyses unless unable to test the dominant leg (i.e., knee replacement) in which case the non-dominant leg will be used.
Total body lean mass | Baseline
  Whole body lean mass will be measured by dual-energy X-ray absorptiometry (DXA).
Appendicular lean mass | Baseline
  Appendicular lean mass will be measured by DXA.
Total body fat mass | Baseline
  Whole body fat mass will be measured by DXA.
Total hip BMD | Baseline
  Bone mineral density (BMD) of the total hip will be measured by DXA.
Femoral neck BMD | Baseline
  Bone mineral density (BMD) of the femoral neck will be measured by DXA.
Lumbar spine BMD | Baseline
  Bone mineral density (BMD) of the lumbar spine (L1-L4) will be measured by DXA.
Subcutaneous abdominal fat | Baseline
  Subcutaneous abdominal fat will be measured by computed tomography (CT).
Visceral abdominal fat | Baseline
  Visceral abdominal fat will be measured by CT.
Thigh inter-muscular adipose tissue | Baseline
  Thigh inter-muscular adipose tissue will be measured by CT.
Glucose | Baseline
  Assessed via a standard clinical assay after fasting for at least 8 hours.
Insulin | Baseline
  Assessed via a standard clinical assay after fasting for at least 8 hours.
Total cholesterol | Baseline
  Assessed via a standard clinical lipid panel after fasting for at least 8 hours
HDL cholesterol | Baseline
  Assessed via a standard clinical lipid panel after fasting for at least 8 hours
LDL cholesterol | Baseline
  Assessed via a standard clinical lipid panel after fasting for at least 8 hours
Triglycerides | Baseline
  Assessed via a standard clinical lipid panel after fasting for at least 8 hours
Systolic blood pressure | Baseline
  Blood pressure will be measured in the right arm using an automated sphygmomanometer with the participant in a seated position after having rested quietly for 10-15 minutes. Participants will sit with feet flat on the floor and legs uncrossed and will be asked not to talk during the rest period or during the measurement. Systolic blood pressure will be defined as the average of three repeated measures.
Diastolic blood pressure | Baseline
  Blood pressure will be measured in the right arm using an automated sphygmomanometer with the participant in a seated position after having rested quietly for 10-15 minutes. Participants will sit with feet flat on the floor and legs uncrossed and will be asked not to talk during the rest period or during the measurement. Diastolic blood pressure will be defined as the average of three repeated measures.
C-reactive protein | Baseline
  C-reactive protein (CRP) will be determined using an automated immunoanalyzer.
Interleukin-6 | Baseline
  Interleukin-6 (IL-6) will be assayed with high-sensitivity Quantikine®.
Soluble tumor necrosis factor receptor 1 | Baseline
  Soluble tumor necrosis factor receptor 1 (sTNFR1) will be assayed with high-sensitivity Quantikine®.

CONTACTS AND LOCATIONS:
Overall Officials: Denise Houston, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States